CLINICAL TRIAL: NCT02508324
Title: Parallel Phase II Trial of IPA Targeted Adoptive Immunotherapy vs Adult Haplo-identical Cell Infusion During Induction of High Risk Leukemia
Brief Title: IPA Targeted Adoptive Immunotherapy vs Adult Haplo-identical Cell Infusion During Induction of High Risk Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual and change in direction of cord blood program
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Blood Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1403014939
Record Dates: First submitted 2015-04-07; First posted 2015-07-24 (Estimated); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cord Blood Unit (Other): The CBU unit must supply a minimum of 0.5 x 10^7/kg and a maximum of 2.5 x 10^7/kg nucleated cell dose pre-cryopreservation. The unit must match at a minimum of 4 of 6 at HLA-A, -B antigens, -DRB1 alleles with the recipient. Mismatches (0-2) can be at any loci. Although molecular level typing will be available for the patient and the CBU unit, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1. The CBU donor will have also undergone HLA typing of the mother, thus allowing determination of the CBU-IPA and NIMA.
  CBU grafts in this study will be investigational units that meet all criteria for clinical use. Better matching units will be preferred over less matching units as long as the CBU dose exceeds 0.5 x 10^7 nucleated blood cells/kg.
  Interventions: Biological: umbilical cord blood unit (CBU)
- Haploidentical (Other): Haploidentical healthy related donor (i.e. parent, child, sibling, possibly third degree or farther removed relative like cousin, aunt, nephew etc.).
  Collected using standard methods and approximately 3 x10^6 CD34 cells/kg will be infused within 72 hours after completion of treatment.
  Interventions: Biological: haplo-identical cells (donor)

INTERVENTIONS:
Biological: haplo-identical cells (donor) — Treatment: Haplo-identical healthy related donor. i.e. Parent, child, sibling, possibly third degree or further removed relative (cousin, aunt, nephew etc). They will be collected using standard methods and approximately 3 x10^6 CD34 cells/kg will be infused within 72 hours after completion of the treatment.
  Arms: Haploidentical
Biological: umbilical cord blood unit (CBU) — Treatment: The CBU unit must supply a minimum of 0.5 x107/kg and a maximum of 2.5x107/kg nucleated cell dose pre-cryopreservation. The unit must match at a minimum of 4 of 6 at HLA-A, -B antigens, -DRB1 alleles with the recipient. Mismatches (0-2) can be at any loci -. Although molecular level typing will be available for the patient and the CBU unit, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1. The CBU donor will also have undergone HLA typing of the mother, thus allowing determination of the CBU-IPA and NIMA. CBU grafts used in this study will be investigational units that meet all criteria for clinical use. Better matching units will be preferred over less matching units as long as the CBU dose exceeds 0.5 x107 nucleated blood cells/kg
  Arms: Cord Blood Unit

SUMMARY:
The purpose of this study is to determine the overall safety of adoptive immunotherapy when given after chemotherapy for AML/MDS. Adoptive immunotherapy means using an infusion of cells from a donor to help fight cancer. The donor cells will be either from the umbilical cord blood (UCB) of a newborn baby or they will be cells collected from a relative (haplo-identical cells).

The 2 cohorts that were discussed - adoptive immunotherapy with either UCB or haplo-identical stem cells - will be analyzed separately.

Preliminary data from other centers has suggested that adoptive immunotherapy with cells from a relative is an effective approach that may improve remission rates and survival in AML and MDS, because they exert anti-cancer effects of their own (so called graft vs leukemia effects) and possibly because they hasten recovery of cell counts from chemotherapy. The Investigators are interested in confirming these data, but also in testing umbilical cord blood cells for the same purpose. Preliminary data indicate that umbilical cord blood cells may have more powerful graft vs leukemia effects and cause fewer side-effects.

DETAILED DESCRIPTION:
This is a phase 2 trial to evaluate the safety of adoptive immunotherapy with Non-Inherited Maternal Antigen (NIMA) compatible, Inherited Paternal Antigen (IPA) targeted CBU or with haplo-identical stem cells after conventional induction therapy for very high risk Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS).

The study has 2 cohorts - patients in cohort 1 will receive CBU cells as adoptive immunotherapy. Patients in cohort 2 will receive haplo-identical cells. Both cohorts will be evaluated separately and no formal statistical comparison between cohorts will be performed.

There will be approximately 20 patients in each cohort, and a 95% confidence interval for the proportion of patients experiencing grade III-IV GVHD complications or unexplained prolonged myelosuppression complications in each cohort can be constructed to be within +/- 13.1% of the observed complication proportions. This calculation assumes an expected prevalence of each of these complication proportions of no greater than 10%.

After 10 patients are enrolled in each group, the incidence of the above-defined life-threatening complications will be assessed. If more than one patient out of 10 enrolled patients (i.e., greater than 10%) in a cohort experiences either of these complications, the cohort will be stopped for safety.

All potential recipients will have complete HLA typing and determination of HLA antibodies. An appropriate umbilical cord blood unit (CBU) will be identified or in the absence of an appropriate CBU, a haplo-identical donor will be identified.

Treatment will be as per the treating physician's choice..

The umbilical cord graft or haplo-graft will be administered between 24 - 72 hours after the completion of the chemotherapy regimen.

The Graft Selection Algorithm is as follows:

1. CBU Unit 5/6 Matched - 1 NIMA match with patient
2. CBU Unit 5/6 Matched - Shared IPA target(s) with patient
3. Haplo-identical relative
4. CBU Unit 4/6 Matched - 1-2 NIMA matches with patient
5. CBU Unit 4/6 Matched - Shared IPA target(s) with patient

Within 42 days of transplant, the recipient's pre-treatment evaluation includes: medical history and physical examinations, Eastern Cooperative Group Oncology Group (ECOG) score, complete blood count (CBC), HLA antibodies, and cytomegalovirus (CMV) antibody testing.

Patients will continue with the therapy specified in this protocol until one of the following occurs:

* Achievement of protocol endpoint complete remission (CR) or CR with incomplete platelet recovery (CRp) after induction and cellular therapy;
* Failure to achieve CR or CRp; or,
* Extraordinary Medical Circumstances: If, at any time the constraints of this protocol are detrimental to the patient's health and/or the patient no longer wishes to continue protocol therapy, remove the patient from protocol treatment. In this event.

After removal from protocol therapy, patients will continue to be followed for survival and disease status. Samples for correlative studies will continue to be collected every two months until one year after cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older
2. Patients with a confirmed diagnosis of AML or MDS, according to World Health Organization (WHO) classification (excluding acute promyelocytic leukaemia) with recurrent or refractory disease as defined below.

   1. For AML:

      1. Primary induction failure (PIF) after ≥ 2 cycles of chemotherapy.
      2. First relapse.
      3. Relapse refractory to salvage chemotherapy
      4. Second or subsequent relapse.
   2. For MDS, either refractory anemia with excess blasts (RAEB) I or RAEB II who failed at least one chemotherapy regimen including either cytarabine or a hypomethylating agent.
3. Patients must have Karnofsky Performance score of ≥70
4. Women of child-bearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to treatment start
5. Patients must be capable of understanding and complying with protocol requirements, and must be able and willing to sign a written informed consent form

Exclusion Criteria:

1. Persistent clinically significant toxicities from previous chemotherapy
2. Known positive status for human immunodeficiency virus (HIV)
3. Pregnant and nursing patients
4. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements
5. Impairment of hepatic or renal function to such an extent that the patient, in the opinion of the investigator, will be exposed to an excessive risk if entered into this clinical study
6. Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure. Any New York Heart Association (NYHA) grade 3 or 4.
7. Any medical condition which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Gomez Arteaga, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Chaekal OK, Scaradavou A, Masson Frenet E, Albano MS, Cushing M, Desai P, Dobrila L, Gergis U, Guarneri D, Hsu JM, Lee S, Mayer SA, Phillips AA, Orfali N, Ritchie EK, Roboz GJ, Romeo C, Samuel MS, Shore T, van Besien K. Adoptive immunotherapy with CB following chemotherapy for patients with refractory myeloid malignancy: chimerism and response. Blood Adv. 2020 Oct 27;4(20):5146-5156. doi: 10.1182/bloodadvances.2020002805. PMID 33091124

RESULTS

PARTICIPANT FLOW:
Groups:
- Cord Blood Unit: The CBU unit must supply a minimum of 0.5 x 10^7/kg and a maximum of 2.5 x 10^7/kg nucleated cell dose pre-cryopreservation. The unit must match at a minimum of 4 of 6 at HLA-A, -B antigens, -DRB1 alleles with the recipient. Mismatches (0-2) can be at any loci. Although molecular level typing will be available for the patient and the CBU unit, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1. The CBU donor will have also undergone HLA typing of the mother, thus allowing determination of the CBU-IPA and NIMA.
  CBU grafts in this study will be investigational units that meet all criteria for clinical use. Better matching units will be preferred over less matching units as long as the CBU dose exceeds 0.5 x 10^7 nucleated blood cells/kg.
  umbilical cord blood unit (CBU): Treatment: The CBU unit must supply a minimum of 0.5 x107/kg and a maximum of 2.5x107/kg nucleated cell dose pre-cryopreservation. The unit must match at a minimum of 4 of 6 at HLA-A, -B antigens, -DRB1 alleles with the recipient. Mismatches (0-2) can be at any loci -. Although molecular level typing will be available for the patient and the CBU unit, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1. The CBU donor will also have undergone HLA typing of the mother, thus allowing determination of the CBU-IPA and NIMA.
- Haploidentical: Haploidentical healthy related donor (i.e. parent, child, sibling, possibly third degree or farther removed relative like cousin, aunt, nephew etc.).
  Collected using standard methods and approximately 3 x10^6 CD34 cells/kg will be infused within 72 hours after completion of treatment.
  haplo-identical cells (donor): Treatment: Haplo-identical healthy related donor. i.e. Parent, child, sibling, possibly third degree or further removed relative (cousin, aunt, nephew etc). They will be collected using standard methods and approximately 3 x10^6 CD34 cells/kg will be infused within 72 hours after completion of the treatment.
Period: Overall Study
Arm/Group | Cord Blood Unit | Haploidentical
Started | 43 | 0
Completed | 43 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled onto the Haploidentical arm due to graft selection criteria and suitable cord blood units being identified for subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cord Blood Unit | Haploidentical | Total
Number analyzed (Participants) | 43 | 0 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 0 | 35
  >=65 years | 8 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 0 | 26
  Male | 17 | 0 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 0 | 7
  Not Hispanic or Latino | 32 | 0 | 32
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 22 | 0 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 43 |  | 43
Primary Malignancy [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia | 39 | 0 | 39
  Myelodysplastic Syndrome | 3 | 0 | 3
  Chronic Myelogenous Leukemia | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of Cellular Immunotherapy as Measured by the Number of Participants Who Developed of Cytokine Release Syndrome (CRS) or Graft-versus-host Disease (GVHD) After Adoptive Immunotherapy
Description: Evaluate the safety of adoptive immunotherapy with Non-Inherited Maternal Antigen (NIMA) compatible, Inherited Paternal Antigen (IPA) targeted CBU or with haplo-identical stem cells after conventional induction therapy for very high risk AML or MDS. Assessed by development of cytokine release syndrome (CRS) or graft-versus-host disease (GVHD) after adoptive immunotherapy.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Unit | Haploidentical
Number analyzed (Participants) | 43 | 0
Participants | 8 | 0

2. Secondary Outcome: Number of Participants Who Developed GVHD by Severity
Description: To assess the incidence and severity of Graft Versus Host Disease (GVHD), after conventional induction therapy followed by adoptive immunotherapy with NIMA compatible, IPA targeted CBU.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Unit | Haploidentical
Number analyzed (Participants) | 43 | 0
Participants
  Grade 1 GVHD | 3 | 0
  Grade 2 GVHD | 0 | 0
  Grade 3 GVHD | 0 | 0
  Grade 4 GVHD | 2 | 0
  No GVHD | 38 | 0

3. Secondary Outcome: Number of Participants With Detectable Cord Blood or Haploidentical Chimerism After Adoptive Immunotherapy
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Unit | Haploidentical
Number analyzed (Participants) | 43 | 0
Participants | 16 | 0

4. Secondary Outcome: Number of Participants With HLA-antibodies That Precluded Them From Moving Forward to Transplant
Description: Count of participants with who developed HLA-antibodies that precluded them from moving forward to transplant
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Unit | Haploidentical
Number analyzed (Participants) | 43 | 0
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Who Responded to Treatment
Description: To assess response rates after adoptive immunotherapy. Response to treatment is defined as effective cytoreduction (ie, <5% residual blasts in a hypocellular bone marrow [BM] or no blasts in an acellular bone marrow [aplasia] obtained ∼14 days after infusion of the CB cells)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Unit | Haploidentical
Number analyzed (Participants) | 43 | 0
Participants | 18 | 0

6. Secondary Outcome: Number of Participants That Underwent a Transplant After Response to Adoptive Immunotherapy
Description: Number of participants that underwent a transplant after response to adoptive immunotherapy. Response to treatment is defined as effective cytoreduction (ie, <5% residual blasts in a hypocellular bone marrow [BM] or no blasts in an acellular bone marrow [aplasia] obtained ∼14 days after infusion of the CB cells)
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cord Blood Unit | Haploidentical
Number analyzed (Participants) | 13 | 0
Participants | 12 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No subjects were enrolled onto the Haploidentical arm due to graft selection criteria and suitable cord blood units being identified for subjects.
Arm/Group | Cord Blood Unit | Haploidentical
All-Cause Mortality (participants affected / at risk) | 5/43 | 0/0
Serious Adverse Events (participants affected / at risk) | 15/43 | 0/0
Other Adverse Events (participants affected / at risk) | 32/43 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cord Blood Unit (N=43) | Haploidentical (N=0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Acute Graft-versus-Host Disease (Investigations) | 3 (3) | 0
Adenovirus Infection (Infections and infestations) | 2 (2) | 0
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0
Fungal Pneumonia (Infections and infestations) | 1 (1) | 0
Fungal sinusitis (Infections and infestations) | 1 (1) | 0
Hypotension (Vascular disorders) | 2 (2) | 0
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0
Multiorgan Failure (Investigations) | 1 (1) | 0
Pneumonia (Infections and infestations) | 1 (1) | 0
Presacral Hematoma (Vascular disorders) | 1 (1) | 0
Post-Transplant Lymphoproliferative Disorder (Investigations) | 1 (1) | 0
Sepsis (Infections and infestations) | 4 (4) | 0
Thromboembolic event (Vascular disorders) | 1 (1) | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cord Blood Unit (N=43) | Haploidentical (N=0)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0
Bacteremia (Infections and infestations) | 18 (19) | 0
BK Viruria (Infections and infestations) | 1 (1) | 0
Enterocolitis Infectious (Infections and infestations) | 7 (7) | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 0
Fungal Pneumonia (Infections and infestations) | 2 (2) | 0
Fungemia (Infections and infestations) | 2 (2) | 0
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0
Pneumonia (Infections and infestations) | 1 (1) | 0
Sinusitis (Infections and infestations) | 1 (1) | 0
Skin Cellulitis (Infections and infestations) | 1 (1) | 0
Thromboembolic Event (Vascular disorders) | 1 (1) | 0
Upper Respiratory Infection (Infections and infestations) | 8 (9) | 0
Urinary Tract Infection (Infections and infestations) | 4 (4) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT02508324/Prot_SAP_000.pdf